CLINICAL TRIAL: NCT05208489
Title: Direct Peritoneal Resuscitation for Intra-abdominal Catastrophes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: New York Medical College (Other)
Responsible Party: Principal Investigator, Kartik Prabhakaran, Trauma Medical Director, New York Medical College
Other Study IDs: 14677
Record Dates: First submitted 2021-12-28; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Intestinal Perforation; Intestinal Obstruction; Trauma Abdomen
MeSH Terms: conditions — Intestinal Perforation; Intestinal Obstruction; Abdominal Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: there is no intervention involved in this study — there is no intervention involved in this study.

SUMMARY:
It is a retrospective study. Patients, who presented with either traumatic or general surgery emergencies, undergone exploratory laparotomy, had an open abdomen management and received Direct Peritoneal Resuscitation in addition to standard resuscitation will be considered as meeting the criteria to collect the data.

DETAILED DESCRIPTION:
Due to the high volume of patient transfers from different facilities with difficult intra-abdominal pathologies and the high case-mix index at Westchester Medical Center, we see many patients who require re-operations and open abdominal management. Since July1st of 2020 we have been using DPR in addition to standard iv fluids on all patients who undergo open abdominal management and it is now standard of care at our facility. we plan to collect the data from all qualified subjects who received DRP since 7/1/2020 to 6/30/2022.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 years of age or older.
* Trauma or General surgery patients who undergo emergency abdominal surgery via laparotomy and who had open abdominal management during the index procedure at our institution.
* Patients who are transferred to our institution with an already open abdomen will also be eligible if they required continued open abdominal management.

Exclusion Criteria:

* Patients <18 years are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients 18 and above, who presents with either traumatic or general surgery emergencies and undergone exploratory laparotomy had an open abdomen management and received DPR in addition to standard resuscitation will be considered as meeting the criteria to be in the study.
Sampling Method: Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2021-12-16 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Post operative outcomes | through out the hospitalization and 30 days after discharge.
  intra abdominal infections and other complications

SECONDARY OUTCOMES:
length of hospital stay | post procedure to 30 days after discharge.
  includes ICU stay, ventilator days and mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Kartik Prabhakaran, MD, Principal Investigator — New York Medical College
Locations (1):
- New York Medical College, Valhalla, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
no plan as of now

REFERENCES:
- [Background] Smith JW, Garrison RN, Matheson PJ, Franklin GA, Harbrecht BG, Richardson JD. Direct peritoneal resuscitation accelerates primary abdominal wall closure after damage control surgery. J Am Coll Surg. 2010 May;210(5):658-64, 664-7. doi: 10.1016/j.jamcollsurg.2010.01.014. PMID 20421025
- [Result] Zakaria el R, Hurt RT, Matheson PJ, Garrison RN. A novel method of peritoneal resuscitation improves organ perfusion after hemorrhagic shock. Am J Surg. 2003 Nov;186(5):443-8. doi: 10.1016/j.amjsurg.2003.07.006. PMID 14599604
- [Result] Crafts TD, Hunsberger EB, Jensen AR, Rescorla FJ, Yoder MC, Markel TA. Direct peritoneal resuscitation improves survival and decreases inflammation after intestinal ischemia and reperfusion injury. J Surg Res. 2015 Dec;199(2):428-34. doi: 10.1016/j.jss.2015.06.031. Epub 2015 Jun 18. PMID 26169030